CLINICAL TRIAL: NCT06257147
Title: A Cluster-randomized Controlled Pragmatic Trial to Evaluate Antimicrobial Stewardship Strategies for Short-course and Oral-switch Antibiotic Therapy for Bloodstream Infections Due to Enterobacterales
Brief Title: Antimicrobial Stewardship for Enterobacterales Bacteremia Management
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Chinese University of Hong Kong (Other)
Responsible Party: Principal Investigator, Grace Lui, Division Head of Infectious Diseases, Department of Medicine & Therapeutics, Chinese University of Hong Kong
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ASP BSI Protocol
Record Dates: First submitted 2024-02-06; First posted 2024-02-13 (Actual); Last update posted 2024-03-20 (Actual); Status verified 2024-03

CONDITIONS: Infections
MeSH Terms: conditions — Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Group 1 wards (physician education) (Placebo Comparator): For Group 1 wards, physician education will be provided. All physicians treating patients in general medical wards will undergo a training session at the start of the study. Education content includes latest evidence on short-course antibiotic therapy and criteria for de-escalation to oral antibiotics for BSI-E. The educational materials will be prepared by Infectious Diseases physicians, and will be presented during one of the monthly departmental meetings, which routinely involve physician education. Ample time will be provided for answering questions from physicians. During the study period, the same material will be presented to new medical staff joining the department. The educational materials will be sent to all physicians in the department regardless of their attendance of the meeting. Patients will receive standard of care.
  Interventions: Behavioral: multifaceted antibiotic stewardship intervention
- Group 2 wards (physician education + paper reminder) (Active Comparator): For Group 2 wards, physician education will be provided as in Group 1. A paper reminder will be attached in the medical records of all consecutive patients on the first working day after Enterobacterale is isolated from blood culture. The reminder documents (1) the clinical and host criteria that should be considered for prescribing short-course antibiotic therapy, and (2) options of oral antibiotics to complete the treatment course. These recommendations are based on results of the trials demonstrating non-inferiority of short-course and oral-switch therapy for BSI-E.
  Interventions: Behavioral: multifaceted antibiotic stewardship intervention
- Group 3 wards (multifaceted antibiotic stewardship intervention) (Active Comparator): Group 3 wards will receive a multifaceted antibiotic stewardship intervention. Physician education will be provided as in Group 1. All consecutive patients fulfilling inclusion and exclusion criteria for study eligibility will be assessed by an Antibiotic Stewardship team. A trained nurse will first assess the patients for clinical and host criteria to determine eligibility for short-course antibiotic therapy. The antibiotic susceptibility test results and the prescribed antibiotics treatment will be reviewed. An Infectious Diseases physician will subsequently make written recommendations for the duration and choice of antibiotic therapy, and provide an appointment within 2 weeks after hospital discharge to review patients' clinical condition when indicated.
  Interventions: Behavioral: multifaceted antibiotic stewardship intervention

INTERVENTIONS:
Behavioral: multifaceted antibiotic stewardship intervention — Group 3 wards will receive a multifaceted antibiotic stewardship intervention. Physician education will be provided as in Group 1. All consecutive patients fulfilling inclusion and exclusion criteria for study eligibility will be assessed by an Antibiotic Stewardship team. A trained nurse will first assess the patients for clinical and host criteria to determine eligibility for short-course antibiotic therapy. The antibiotic susceptibility test results and the prescribed antibiotics treatment will be reviewed. An Infectious Diseases physician will subsequently make written recommendations for the duration and choice of antibiotic therapy, and provide an appointment within 2 weeks after hospital discharge to review patients' clinical condition when indicated.

SUMMARY:
We hypothesize that a multifaceted antibiotic stewardship intervention incorporating physician education, prospective chart review with antibiotic recommendation, and provision of follow-up by a multidisciplinary antibiotic stewardship team, is more effective than physician education and reminders alone in improving physicians' prescription of short-course and oral-switch antibiotic therapy for patients with bloodstream infections due to Enterobacterales (BSI-E).

This study is to:

1. determine the effectiveness of a multifaceted antibiotic stewardship intervention in improving physicians' prescription of short-course antibiotic therapy for BSI-E
2. determine the effectiveness of a multifaceted antibiotic stewardship intervention in improving physicians' de-escalation to oral antibiotic therapy for BSI-E

DETAILED DESCRIPTION:
Antimicrobial resistance is a major global threat, causing 5 million deaths globally in 2019. One of the crucial strategies to control the emergence and spread of multidrug-resistant organisms (MDRO) is to minimize unnecessary antibiotics exposure.

Shorter duration of antibiotic therapy and oral-switch therapy for bloodstream infection due to Enterobacterales (BSI-E) had demonstrated similar treatment success and clinical outcomes as compared with longer courses in randomized controlled trials. Despite the release of such data, clinicians may be reluctant to shortern duration of therapy for BSI-E and adopt oral-switch approach.

This study aims to determine the optimal approach to aid clinicians in adopting evidence-based practice in a clinical setting. This study is a pragmatic cluster-randomized controlled trial in the medical wards of an acute hospital. A cluster, as the unit of randomization, is a medical ward. Medical wards will be randomized to three groups: (1) physician education only; (2) physician education and paper reminder; (3) multifaceted antibiotic stewardship intervention. The prescription of antibiotic therapy by treating physicians and outcomes of patients with BSI-E will be studied.

Patients' antibiotics regimen and clinical outcomes in the three groups will be compared.

ELIGIBILITY:
Inclusion Criteria:

* aged ≥18 years;
* hospitalization in one of the medical wards of the hospital; and
* isolation of Enterobacterales in at least one blood culture bottle, where Enterobacterales include Escherichia coli, Klebsiella, Proteus, Enterobacter, Serratia, Citrobacter, Providencia and Morganella species.

Exclusion Criteria:

* concomitant isolation of pathogens other than Enterobacterales in blood or other relevant clinical specimens;
* infections requiring prolonged courses of antibiotics, such as intra-abdominal abscess, central nervous system infection, endocarditis, lung abscess or empyema, osteomyelitis, and prostatitis;
* focus of infection not controlled;
* nosocomial infection with onset within 7 days; or
* Presence of neutropenia, allogenic stem cell transplant within one year, use of high-dose steroid (>40mg prednisolone or equivalent for > 2 weeks), or
* died before day 7 will be excluded from the analysis, or
* already on more than 7 days of antibiotics for BSI-E at the time of screening.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 420 (Estimated)
Dates: Start 2024-05-01 (Estimated); Primary Completion 2026-11-30 (Estimated); Study Completion 2026-11-30 (Estimated)

PRIMARY OUTCOMES:
Percentage of patients receiving 7 days effective antibiotic therapy for the treatment of BSI-E | 7 days
  proportion of patients receiving 7 days of effective antibiotic therapy for the treatment of BSI-E

SECONDARY OUTCOMES:
proportion of patients with susceptible oral antibiotics completed the course with an oral antibiotic | during hopsitalization
  proportion of patients with susceptible oral antibiotics completed the course with an oral antibiotic
30-day all-cause mortality | 30 day since hospital admission
  30-day all-cause mortality
clinical failure | within 90 days since hopsitalization
  clinical failure , defined as relapse of BSI-E due to the same Enterobacterales, local suppurative complications or distant complications due to the same pathogen within 90 days
length of stay in hospital | from the admission up to the discharge
  length of stay in hospital
re-admission to hospital within 90 days | within 90 days since discharge
  re-admission to hospital within 90 days

CONTACTS AND LOCATIONS:
Locations (1):
- Prince of Wales Hospital, Shatin, Hong Kong

IPD SHARING:
Plan to Share IPD: No